CLINICAL TRIAL: NCT07137143
Title: The Effect of Heating the Intensive Care Room in the Early Postoperative Period on Patient Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Cansel Bozer, expert, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CU-SBF-CB-05
Record Dates: First submitted 2025-08-16; First posted 2025-08-22 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Abdominal Surgery Complications; Hypothermia Following Anesthesia
Keywords: intensive care unit; hypothermia; postoperative warming
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Intervention Model Description: 2 groups, control group and intervention group
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- no intervention group (No Intervention): In the preoperative period, patients with a body temperature of 36°C-37°C one hour before surgery will be included in the sample. Postoperatively, upon arrival from the operating room to the intensive care unit, which has a humidity range of 55%-65% and a temperature range of 22°C-25°C, will be safely transferred to a single-bed room, monitored, and wiped down. After ensuring personal hygiene, the patient will be covered with a 160x220cm cotton quilt. The heating device hose will be placed inside the bed from the side of the bed. The electric heater will be operated at 38°C (Medium) for 120 minutes, 15 cm from the patient's body. Routine treatment and care will then be administered. Vital signs, shivering level, and temperature perception will be recorded on the patient's follow-up form at 0, 15, 30, 45, 60, 90, and 120 minutes postoperatively.
- intervention group (Experimental): In the preoperative period, patients with a body temperature of 36°C to 37°C one hour before surgery will be included in the sample. In the postoperative period, the intensive care room, which has a routine humidity range of 55%-65% and a temperature of 22°C to 25°C, will be heated to the upper limit of the intensive care room temperature range, 27°C, with an electric heater half an hour before the operation. After ensuring personal hygiene, the patient will be safely transferred to the bed in the single room, monitored, and wiped down. After ensuring personal hygiene, the patient will be covered with a 160x220cm cotton quilt. The heating device hose will be placed inside the bed from the edge of the bed. The electric heater will be operated at 38°C (Medium Level) for 120 minutes, 15cm from the patient's body. Routine treatment and maintenance will be administered. Then, the vital signs, pain, shivering level, and temperature perception will be recorded in the patient follow-up form a
  Interventions: Other: The rooms of the intervention group patients will be heated before they come to intensive care and the temperature of the room will be increased.

INTERVENTIONS:
Other: The rooms of the intervention group patients will be heated before they come to intensive care and the temperature of the room will be increased. — The rooms of the intervention group patients will be heated before they come to intensive care and the temperature of the room will be increased.
  Arms: intervention group

SUMMARY:
The aim of this study was to evaluate the effect of heating the intensive care room in the early postoperative period on patient outcomes.

DETAILED DESCRIPTION:
Hypothermia is defined as a drop in body temperature below 35°C, and patients are at high risk during the perioperative period.Unintentional hypothermia can begin before anesthesia and continue for up to the first 24 hours postoperatively.Its incidence varies between 50% and 90% depending on the patient's medical condition, the nature of the surgery, and operating room conditions.Hypothermia leads to complications such as arrhythmia, hypertension, angina, coagulopathy, increased oxygen demand, nausea, vomiting, and delayed wound healing.Additionally, adverse effects such as shivering, changes in cognitive function, decreased patient comfort, and prolonged hospital stay are also observed.The development of hypothermia is influenced by anesthesia-related thermoregulation impairment, a cold operating room environment, and prolonged operations.Patients report experiencing intense chills and shivering, especially in the postoperative period.

This increases anxiety and negatively impacts patient satisfaction and comfort. Guidelines recommend the use of passive and active warming methods to prevent unintended hypothermia.However, no studies have been found in the literature examining the effect of heating the patient room in the postoperative period.In this regard, our study was designed to evaluate the effect of heating the intensive care room in the early postoperative period on patient outcomes and to contribute to the literature.

ELIGIBILITY:
Inclusion Criteria:

* The following criteria will be included in the sample:
* Patients who underwent elective abdominal surgery and were admitted to intensive care after surgery.
* Patients aged 18 and over.
* Patients whose body temperature on the morning of surgery was neither below 36°C nor above 37.5°C.
* Patients who did not have a pacemaker, dementia, advanced spasticity, muscle atrophy, peripheral lesions, osteoporosis, skin irritation, diabetes, hypertension, or obesity.
* Patients who did not require mechanical ventilation.
* Patients who did not have any illness that would impair thermoregulation (such as head trauma or hypothalamic damage).

  • Patients who were not taking medications that would affect thermoregulation, such as vasodilators.
* Patients who did not have peripheral circulation problems.
* Patients who were not alcohol or substance abusers.
* Patients who did not have mental retardation.
* Patients who were conscious and oriented to person, time, and place.
* Patients who could speak Turkish.
* Patients who did not have any auditory or visual impairments.
* Patients who volunteered for the study.

Exclusion Criteria:

* Patients who do not meet the sampling criteria, who develop postoperative complications (bleeding, intubation, stenosis, necrosis, ileus, dermatitis, parastomal herniation, etc.), and whose relatives do not consent to the study will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-04-20 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
The Thermal Comfort Scale (TKS) | 6 months
  The Thermal Comfort Scale (TKS) is a Likert-type scale developed by Wagner and colleagues in 2006. Although it was developed to assess the thermal comfort perception of preoperative patients, the authors state that it is also suitable for evaluating conscious postoperative patients. The scale assesses the patient's thermal comfort perception based on self-report. The scale consists of 13 items, each scored from 1 to 6. A higher score indicates a higher thermal comfort perception.
Temperature Comfort Perception Scale (TPS) | 6 months
  The Temperature Comfort Perception Scale is a visual analog scale developed by Wagner and colleagues to objectively assess patients' perception of temperature comfort. It is scored based on patient self-reporting from 0 (extremely cold) to 10 (extremely hot), with a score of 5 representing optimal temperature comfort.
Numerical Pain Assessment Scale (SAS) | 6 months
  This study planned to use a 10-point pain scale, with 0 representing no pain and 10 representing the most unbearable pain. In the study, patients will be asked to select the number that best describes their pain intensity.
Tremor Level Assessment Scale (TRS) | 6 months
  Tremor Level Assessment Scale (TRS) This form, used to assess patients' tremor levels, was developed based on literature. The form was developed using the studies of Badjaita et al. (2008) and May et al. (2011), and was based on criteria for determining the level of tremor based on observation. Tremor level will be assessed based on observation as follows: 0 (absent), 1 (mild; tremor localized only to the neck and/or thorax), 2 (moderate; tremor in the neck, thorax, and upper extremities), and 3 (severe; tremor in the trunk, upper, and lower extremities).
Patient Monitoring Form (PMP) | 6 months
  Patient Monitoring Form (PMP) This form was developed by researchers based on a literature review to monitor the body temperature, blood pressure, pulse, respiration, pain, oxygen saturation, shivering levels, thermal comfort perception, and thermal comfort levels of patients in the intervention and control groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Adana City Training and Research Hospital, Adana, Yüreğir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No